CLINICAL TRIAL: NCT00753623
Title: Clinical Management of Neuropathic Pain With Ramelteon
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment did not accrue as expected.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Principal Investigator, Jianren Mao, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008P-000988
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Results first posted 2014-07-18 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Neuropathic Pain
Keywords: Pain; Neuropathic pain; Pain scores
MeSH Terms: conditions — Neuralgia; Pain | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ramelteon first, placebo second (Active Comparator): In a crossover design, a subject will be first assigned to the ramelteon arm and then switched over to the placebo arm. As this is a double-blind study, neither the subject nor the study staff will know which intervention the subject is randomly assigned. The ramelteon dose is 8mg once a night.The ramelteon and placebo will be blinded by the central pharmacy.
  The subject is randomly assigned to first receive either ramelteon or placebo. The first intervention will be 14 days long. There is a 7 day washout period, and then the subject is assigned to the opposite intervention. The second intervention will be 14 days long.
  Interventions: Drug: Ramelteon; Drug: Placebo
- Placebo first, ramelteon second (Placebo Comparator): In a crossover design, a subject will be first assigned to the placebo arm and then switched over to the ramelteon arm. As this is a double-blind study, neither the subject nor the study staff will know which intervention the subject is randomly assigned. The ramelteon dose is 8mg once a night. The ramelteon and placebo will be blinded by the central pharmacy.
  The subject is randomly assigned to first receive either ramelteon or placebo. The first intervention will be 14 days long. There is a 7 day washout period, and then the subject is assigned to the opposite intervention. The second intervention will be 14 days long.
  Interventions: Drug: Ramelteon; Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon — ramelteon (8 mg)
  Other Names: Rozerem
Drug: Placebo — In a crossover design, a subject will be first assigned to the ramelteon or placebo arm and then switched over to the opposite arm.

SUMMARY:
This proposal is to conduct a double-blinded, randomized, placebo-controlled, crossover clinical study to examine the hypothesis that ramelteon would reduce pain score and improve functional status in subjects with neuropathic pain.

DETAILED DESCRIPTION:
Neuropathic pain is a chronic pain condition resulting from injury to the peripheral and/or central nervous system. Despite extensive research over the last several decades, neuropathic pain remains poorly managed due to the lack of effective pharmacological tools. To date, little has been known regarding the effect of melatonin and its analogues on clinical neuropathic pain. We propose to conduct a randomized, placebo-controlled, double-blinded, and crossover clinical trial to examine the effect of ramelteon [a melatonin (MT) 1/ MT2 receptor agonist] on neuropathic pain. We hypothesize that ramelteon would reduce pain score and improve functional status in subjects with neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

1. Subject will be between ages 18 to 65 years.
2. Subject has not been on ramelteon for at least one month.
3. Subject agrees to make no change in his/her current pain medications during the entire study period (5 weeks). This requirement will ensure that valid comparisons of primary and secondary measures can be made before and after the study.
4. Subject has a VAS pain score of 5 or above at the beginning of the study.
5. Subject has had a neuropathic pain condition as listed above for at least three months. This requirement is to avoid clinical uncertainty from an unstable pain condition and to minimize the study variation.
6. Female subjects of childbearing potential must have a negative urine pregnancy test at the initial visit.

Exclusion Criteria:

1. Subject has moderate to severe liver impairment.
2. Subject has Liver Function Tests (LFT's) >1.5X normal.
3. Subject has a history of renal impairment.
4. Subject has moderate or severe cardiac or pulmonary disease including a base line oxygen saturation of less than 95% on room air or any requirement for supplemental oxygen.
5. Subject has a history of glaucoma.
6. Subject has obstructive sleep apnea.
7. Subject is taking medications for sleep disorders including insomnia.
8. Subject has a major psychiatric disorder (major depression requiring a recent hospitalization within three months prior to the study; bipolar disorder; schizophrenia; psychotic disorders; substance abuse).
9. Subject has a history of dementia or delirium.
10. Subject has a history of falls.
11. Subject is pregnant or lactating.
12. Subject is using an illicit drug detected by a screening test.
13. Subject is currently taking Fluvoxamine.
14. Subject has been taking Ketoconazole in the past two weeks.
15. Subject has known hypersensitivity to ramelteon.
16. Subject has pending litigation related to his/her neuropathic pain condition.
17. Subject has Concurrent participation in other research drug trials or other study participation within 30 days of enrollment in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-09; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jianren Mao, M.D., Ph. D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in person at the MGH Center for Pain or by advertisement throughout MGH and the local community.
Groups:
- Placebo Phase I; Ramelteon Phase II: In a crossover design, a subject was first assigned to the placebo and then switched over to the ramelteon.
  Ramelteon : ramelteon (8 mg)
- Ramelton Phase I; Placebo Phase II: In a crossover design, a subject was first assigned to the ramelteon and then switched over to the placebo.
  Ramelteon : ramelteon (8 mg)
Period: Phase I (14 Days)
Arm/Group | Placebo Phase I; Ramelteon Phase II | Ramelton Phase I; Placebo Phase II
Started | 11 | 12
Completed | 9 | 8
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Physician Decision | 1 | 2
Not completed — Adverse Event | 0 | 1
Period: Washout (7 Days)
Arm/Group | Placebo Phase I; Ramelteon Phase II | Ramelton Phase I; Placebo Phase II
Started | 9 | 8
Completed | 8 | 8
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0
Period: Phase II (14 Days)
Arm/Group | Placebo Phase I; Ramelteon Phase II | Ramelton Phase I; Placebo Phase II
Started | 8 | 8
Completed | 8 | 7
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Phase I; Ramelteon Phase II | Ramelton Phase I; Placebo Phase II | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 23
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 4 | 7 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Difference in Visual Analog Scale (VAS) for Pain (0-10) Between Treatments
Description: Subjects were asked to rate their pain the VAS with 0 being no pain and 10 being the worst pain they can imagine. The VAS scores were compared between the baseline and after a period of treatment. A negative number indicates an improvement in pain from baseline score.
Time Frame: VAS score at baseline and after the treatment period
Population: Only 15 subjects completed both treatment phases so we only included these subjects in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ramelteon: Participants who received Ramelteon 8 mg during the first or last 2 weeks of the study.
- Placebo: Participants who received placebo medication during the first or last 2 weeks of the study.
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 15 | 15
units on a scale | -1.0 (1.4) | -1.1 (1.5)
Statistical Analysis 1: Comparison: Ramelteon vs Placebo; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Two weeks for each intervention and a 1 week period of no intervention in between phases.
Arm/Group | Ramelteon | Placebo
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramelteon (N=23) | Placebo (N=23)
Hospitalization (Immune system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Problems with recruitment and termination of the study consequently resulted in uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No